CLINICAL TRIAL: NCT00745017
Title: Stress Generation and Recurrent Depression: The Role of Differential Treatment Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Kate Leslie Harkness, PhD, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091/2003
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Last update posted 2008-09-01 (Estimated); Status verified 2008-08

CONDITIONS: Depression; Major Depressive Disorder
Keywords: recurrent depression; major depressive disorder; interpersonal therapy; cognitive behavioral therapy; antidepressant therapies; outome predictors; personality dimensions
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (Experimental)
  Interventions: Behavioral: Interpersonal Therapy
- 3 (Experimental)
  Interventions: Drug: Antidepressant medication

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — All patients randomized to this condition will receive 16 consecutive weeks of manualized cognitive-behaviour therapy provided by either M.S.W or Ph.D. psychotherapists trained and certified in CBT. Treatment will be conducted according to the manualized CBT treatment for depression outlined by Beck and colleagues (Beck et al., 1979), and consistent with the protocol administered in the NIMH study.
  Arms: 1
Behavioral: Interpersonal Therapy — All patients randomized to this condition will receive 16 consecutive weeks of manualized interpersonal psychotherapy conducted by M.S.W., Ph.D., or M.Ed. psychotherapists trained and certified in IPT.
  Arms: 2
Drug: Antidepressant medication — Patients patients randomized to this condition will be treated for 16 weeks with different classes of anti-depressant medications, using standardized protocols. Patients will receive 16 weeks of treatment with either a SSRI (sertraline or paroxetine) or a SNRI (venlafaxine). The dose range is as follows: sertraline 50-200 mg/day, paroxetine 20-40 mg/day, venlafaxine 75-375 mg/day. Patients unable to continue with the prescribed medication due to side effects and/or lack of response will be prescribed an alternate medication during the first two weeks of the protocol.
  Arms: 3

SUMMARY:
Depression affects over one million people in Canada, resulting in $14.4 billion per year in costs to Canadian society. In order to prevent this often lifelong disorder, it is critically important to identify risk factors for the recurrence of depression. A crucial force in maintaining depression is the generation of stressful life events. That is, individuals who have a history of depression are likely to generate the very events that precipitate future depressive episodes (e.g., relationship break-up, fired from job, conflicts with the law) due to negative personality characteristics and disrupted social support networks resulting from previous episodes. This project is the first to test a model that examines the role of negative personality, low social support, and childhood abuse and neglect as risk factors for the generation of stressful life events that predict future depression. We will test this model in a group of patients meeting formal criteria for depression who will be treated and then followed up for 12 months or until depression recurrence. With this long-term design we will be in a unique position to understand how depression is maintained over time, thus suggesting important treatment strategies to prevent depression recurrence.

DETAILED DESCRIPTION:
The National Institute of Mental Health (NIMH) Treatment of Depression Collaborative Research Programme (TDCRP) (Elkin et al., 1989; Sotsky et al., 1991) compared three forms of treatment for depression -- imipramine plus clinical management (IMI-CM), cognitive behaviour therapy alone (CBT), interpersonal therapy alone (IPT) -- against a placebo control plus clinical management (PLA-CM) condition. These three treatments were found equally effective in the treatment of the index episode of depression when compared to the placebo control (Elkin et al., 1989). The results from the TDCRP study also indicated that patient characteristics, irrespective of treatment modality, were predictive of treatment effects. Six patient dimensions -- social dysfunction, cognitive dysfunction, expectation for improvement, endogenous features, double depression and duration of current episode -- were all found to be significant predictors of outcome (Sotsky et al., 1991). Patient characteristics were also found to be associated with differential outcome depending on treatment modality. Elevated social dysfunction, for example, interfered with successful outcome in IPT, whereas cognitive dysfunction hindered successful outcome with CBT. Cognitive dysfunction also predicted poor treatment response in the IMI-CM condition. Cognitive vulnerability would be expected to mediate response to treatment in CBT, as the presumed mechanism of change is dysfunctional depressogenic cognitions (e.g., Beck et al., 1979; Whisman, 1993). The finding that cognitive vulnerability was also implicated in treatment response to a pharmacological intervention is without theoretical explanation or specific causal agency.

The purpose of the proposed research is to further examine the relationship between treatment outcome and patient characteristics associated depression. In particular, the relationship between treatment outcome and two personality/cognitive characteristics implicated as vulnerability factors for depression - self-criticism and dependency - will be explored.

The first aim of the proposed investigation is to examine the relationship between change in self-criticism and dependency and the relationship of this change to treatment response and reduction in severity of depression. Mode-specific outcome measures will be administered to outpatients with major depression randomly assigned and treated with CBT, IPT or PHT.

The second aim of this study is to examine the issue of whether successful targeting of either cognitive dysfunction in CBT or interpersonal functioning in IPT will result in a reduced risk for relapse and/or recurrence of a major depressive episode.

We believe that the dependent type, who centres their definition of self entirely around issues of affiliation with others, would be more likely to show changes related to such themes in a therapeutic intervention specifically designed to address interpersonal problems. In contrast, the self-critic who defines self primarily around issues related to achievement and engages in excessively harsh and unrealistic self-appraisal would respond best to an intervention that targeted these punitive cognitions.

HYPOTHESES/RESEARCH QUESTIONS

Prediction of Treatment Outcome (Objective 1):

Two sets of hypotheses are proposed. In all analyses the DEQ will be used to assess self-criticism and dependency. The first set of hypotheses involves mode specific treatment outcomes and the second set of hypotheses address differences in the mechanisms of change across the treatments.

The first set of hypotheses are: (a) all treatments will be equally effective in the treatment of the index episode, (b) baseline self-criticism and dependency scores will predict outcome in all treatments, with higher self-criticism and dependency scores related to poor outcome, (c) CBT will demonstrate greater specificity for targeting self-criticism than will either PHT or IPT, (d) IPT will demonstrate greater specificity for treating interpersonal functioning than will either PHT or CBT, (e) PHT will demonstrate greater specificity for treating endogenous symptoms than will either CBT or IPT.

The second set of hypotheses are: (a) change in self-criticism scores and dysfunctional cognitions will mediate a positive treatment response in CBT but not in IPT or PHT, (b) change in dependency scores and interpersonal deficits will mediate positive treatment response in IPT but not in CBT or PHT, (c) change in endogeneity will mediate positive treatment response in PHT but not in CBT or IPT.

Prediction of Relapse and Recurrence (Objective 2):

It is hypothesized that: (a) CBT and IPT will produce a lower rate of relapse and recurrence than PHT because of the greater reduction in stable dysfunctional cognitions related to either self-critical and/or interpersonal vulnerabilities; (b) in cases where interpersonal vulnerabilities are predominant, IPT will produce lower rates of relapse and recurrence than either CBT and PHT, in cases where self-critical vulnerabilities are predominant, CBT will produce lower rates of relapse and recurrence than either IPT or PHT.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for DSM-IV diagnosis of non-psychotic, major depression based on the Structured Interview for DSM-IV, Axis I disorders
* Score > 16 the 17-item Hamilton Rating Scale for Depression
* Ages between 18 and 60
* Are medication-free (i.e., of antidepressants) for a minimum of two weeks prior to treatment are eligible for entry into treatment protocols
* Minimum eight grade education and fluency in reading English
* Ability to give informed consent and complete assessment instruments unassisted

Exclusion Criteria:

* a SCID-I diagnosis of:

  * Bipolar Disorder (past or present),
  * Schizoaffective Disorder,
  * Schizophrenia,
  * Substance Abuse Disorder (current or within the past 6 months),
  * Borderline or Antisocial Personality Disorder,
  * Organic Brain Syndrome
* Electroconvulsive Therapy (ECT) within the past 6 months
* Concurrent active medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2001-07; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: Kate L Harkness, PhD, Principal Investigator — Queen's University
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada